CLINICAL TRIAL: NCT02063061
Title: Low-energy Linear Extracorporal Shock Wave Therapy for Erectile Dysfunction.
Acronym: ESWTvsED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grzegorz Fojecki (Other)
Collaborators: University of Southern Denmark (Other); Region of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Grzegorz Fojecki, MD, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIV-13-07-011546
Record Dates: First submitted 2014-01-09; First posted 2014-02-14 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Erectile Dysfunction
Keywords: extracorporeal shock wave therapy ESWT; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham treatment (Sham Comparator): Subject will answer standardized questionnaires. Sham treatment arm will receive initially 5 sham series and after they answer standardized questionnaires they will receive 5 series of active treatment. Afterwards patients will answer standardized questionnaires again.
  Interventions: Device: Sham treatment; Device: ESWT treatment
- ESWT treatment (Active Comparator): Subject will answer standardized questionnaires. Subjects will receive 10 treatments with ESWT. Afterwards patients will answer standardized questionnaires again.
  Interventions: Device: ESWT treatment

INTERVENTIONS:
Device: Sham treatment — Patients will receive simulated treatment, with the same ESWT unit as in other arm. Placebo gel-pad is design to prevent shockwaves emission. Looks identical as active gel-pad.
  Other Names: Sham
  Arms: Sham treatment
Device: ESWT treatment — ESWT treatment group will receive 600 low-energy, linear shockwaves against erectile dysfunction per week in 10 weeks.
  Other Names: ESWT

SUMMARY:
The purpose of this study is to determine whether extracorporeal shock wave therapy (ESWT) is an effective treatment for erectile dysfunction.

DETAILED DESCRIPTION:
Erectile dysfunction has a negative impact on quality of life and relationships. Thirty to sixty- five percent of men over 40 years of age have erection disorders. Current challenges of medical treatment are met with high costs and risks of side effects. Emerging new therapy with low-energy shock waves stimulate production of endothelial growth factor and nitrogen oxide which results in angiogenesis. It is our aim to assess efficaciousness of this method on potential to improve erectile dysfunction. We propose a prospective double-blind, randomised, cross-over, sham-controlled trial, to assess how effective shock waves therapy is for erectile dysfunction. Patients will receive one treatment per week for ten weeks. Subjects will be followed for up to one year after treatment. Standardized questionnaires will assess study endpoints for erectile dysfunction. We hypothesize that shock wave therapy could represent a low cost, low risk treatment for erectile dysfunction in men.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction for at least 6 months
* In relationships
* Patient accept not to use any other therapy against erectile dysfunction

Exclusion Criteria:

* Prostatectomy
* Radiotherapy in pelvis
* Hormonal therapy against prostate cancer
* Anatomical penis disorder
* Penile prosthesis
* Treatment with anticoagulants (except acetylsalicylic acid 75 mg)
* Psychiatric disorder
* Hypogonadism
* IIEF score higher than 25
* Pregnant partner og delivered within last 12 months
* Critical health disease
* Neurological disorders

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) outcome increases by 5 points | 1 year

SECONDARY OUTCOMES:
Erectile Hardness Scale (EHS) outcome is equal or higher than 3. | 1 year

OTHER OUTCOMES:
Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) outcome | 18 weeks
  Assesed after complition af clinical trial
Number of Participants with Adverse Events | 18 weeks
  During treatment period all patients will be examined for advers events

CONTACTS AND LOCATIONS:
Overall Officials: Palle Oshter, professor, Study Director — University of Southern Denmark
Locations (1):
- Hospital of Southern Denmark, Sønderborg, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gruenwald I, Appel B, Kitrey ND, Vardi Y. Shockwave treatment of erectile dysfunction. Ther Adv Urol. 2013 Apr;5(2):95-9. doi: 10.1177/1756287212470696. PMID 23554844
- [Result] Gruenwald I, Appel B, Vardi Y. Low-intensity extracorporeal shock wave therapy--a novel effective treatment for erectile dysfunction in severe ED patients who respond poorly to PDE5 inhibitor therapy. J Sex Med. 2012 Jan;9(1):259-64. doi: 10.1111/j.1743-6109.2011.02498.x. Epub 2011 Oct 18. PMID 22008059
- [Result] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- See also: regional ethical committee — http://komite.regionsyddanmark.dk/wm258128
- See also: University of Southern Denmark — http://www.sdu.dk/